CLINICAL TRIAL: NCT00950196
Title: The Effect of Amantadine on Movement Disorder in Ataxia-Telangiectasia
Brief Title: Amantadine for Improving Neurologic Symptoms in Ataxia-Telangiectasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Andreea Nissenkorn, MD, Pediatric Neurologist, Director National A-T Clinic, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-08-5196-AN-CTIL
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Ataxia; Chorea; Dystonia; Parkinsonism; Fatigue
MeSH Terms: conditions — Ataxia; Chorea; Dystonia; Parkinsonian Disorders; Fatigue | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- amantadine (PKMERZ) (Experimental)
  Interventions: Drug: amantadine sulphate

INTERVENTIONS:
Drug: amantadine sulphate — amantadine 5/mg/kg for 2 month- tapered up during 2 weeks at 1 month possibility to increase dosage to 8 mg/kg or reduce it if there are side effects
  Other Names: PKMERZ

SUMMARY:
Ataxia-Telangiectasia A-T is a neurodegenerative disorder of the cerebellum, manifesting with ataxia, as well as extrapyramidal features. Treatment of A-T is discouraging, since no treatment seems to change the course of disease, but improvement can be achieved by symptomatic treatment of the bothersome movement disorder . While various dopaminergic agents are occasionally used, reports of benefit are rather sparse and anecdotal. Amantadine, a well known drug used in influenza as well as movement disorder of Parkinson, has been proved to improve various other types of movement disorder as ataxia, chorea, dystonia, akinesia and attention span. The purpose of this study is to investigate weather amantadine sulphate improves ataxia and the movement disorder (bradykinesia, parkinsonism, dystonia, chorea), as well as the general well being in patients with A-T.

DETAILED DESCRIPTION:
Ataxia-Telangiectasia (A-T) is a complex multisystem disorder with neurodegenerative course, immune deficiency, and tendency to develop malignancies .The clinical picture includes progressive cerebellar ataxia along with a movement disorder (chorea, dystonia or bradykinesia) that may be even more disabling than the ataxia . Fatigability, drooling and reduced stamina are other major concerns. Disease course is devastating: towards the second decade of life the affected children are usually bound to wheelchair and survival beyond the second decade of life is rare. Treatment of A-T is discouraging, since no treatment seems to change the course of disease, but improvement can be achieved by symptomatic treatment of the bothersome movement disorder . While various dopaminergic agents are occasionally used, reports of benefit are rather sparse and anecdotal.

Amantadine is a dopaminergic agent approved for prophylaxis of influenza (in children over 1 year of age and adults) as well as for extrapyramidal disorders in adults: Parkinson disease and drug induced dyskinesias . Amantadine increases dopaminergic transmission by inhibiting its synaptic uptake, as well as an antagonizing the striatal NMDA receptors). Additional conditions found to be improved with amantadine are: cerebellar ataxia, vigilance after brain trauma in adults and children ,attention deficit disorder in children, chorea and akinesia in Huntington's disease .

Amantadine is an FDA approved drug for treatment and prevention of influenza, Parkinson disease and drug induced dyskinesia; it is approved for use in adults and children over 1 year of age.

Dosage in children: 5 mg/kg body weight up to 8.8mg/kg/. Dosage in adults: 200 to 300 mg/day. The daily dosage should be divided into 2 to 3 daily portions. Amantadine is a safe drug with mild side effects: headache, decreased appetite, sedation, fatigue, abdominal pain, vomiting, insomnia, pedal edema and rash (4-10).

Studies in children proved amantadine to be a safe and tolerable drug. Amantadine was administered to 24 healthy children with ADHD, aged 5-13 year old . Side effects were present in 13/24 and were usually mild: decreased appetite, headache, sedation, mild insomnia, vomiting, fatigue, abdominal pain. One subject dropped out because of headache. Six low response children after traumatic brain injury were treated with amantadine (concurrently with other medication) The drug was safe with relatively mild side effects: sedation, intermittent tremor, dizziness, but no serious side effects requiring discontinuation of the protocol.

Study purpose The purpose of this study is to investigate weather amantadine sulphate improves ataxia and the movement disorder (bradykinesia, parkinsonism, dystonia, chorea), as well as the general well being in patients with A-T.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of A-T
* significant functional disability
* age over 4 years

Exclusion Criteria:

* major comorbidity: active malignancy requiring chemotherapy, kidney or liver failure
* sexually active
* known hypersensitivity to amantadine
* previous treatment with amantadine in the 2 months preceding the study

Ages: 4 Years to 50 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
improvement in ataxia | 2 month

SECONDARY OUTCOMES:
improvement in extrapyramidal movement disorder | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Nissenkorn, MD, Principal Investigator — Sheba Medical Center, Pediatric Neurology and National A-T Clinic
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Nissenkorn A, Hassin-Baer S, Lerman SF, Levi YB, Tzadok M, Ben-Zeev B. Movement disorder in ataxia-telangiectasia: treatment with amantadine sulfate. J Child Neurol. 2013 Feb;28(2):155-60. doi: 10.1177/0883073812441999. Epub 2012 May 1. PMID 22550086